CLINICAL TRIAL: NCT03562494
Title: A Randomized, Sham Surgery Controlled, Double-blind, Multi-center, Phase 1 Clinical Trial, Evaluating the Safety of VY-AADC02 in Moderate to Advanced Parkinson's Disease Patients With Motor Fluctuations
Brief Title: VY-AADC02 for Parkinson's Disease With Motor Fluctuations (RESTORE-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Voyager Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PD-1105
Record Dates: First submitted 2018-05-16; First posted 2018-06-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease (PD); Aromatic L-Amino Acid Decarboxylase; AADC; AAV; VY-AADC02; AAV2-hAADC; DDC; Gene Therapy; Levodopa; Dopamine; Neurosurgery; NBIb-1817; Motor Fluctuations
MeSH Terms: conditions — Parkinson Disease | interventions — salicylhydroxamic acid; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomized, Sham Surgery Controlled, Double-blind, Multi-center
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VY-AADC02 (NBIb-1817) (Experimental): Single administration of up to 3.6 x 10^12 vector genomes (vg) of VY-AADC02
  Interventions: Biological: VY-AADC02
- Sham (Placebo) Surgery (Placebo Comparator): Sham surgical procedure
  Interventions: Other: Sham (Placebo) Surgery

INTERVENTIONS:
Biological: VY-AADC02 — Adeno-associated viral vector serotype 2 encoding human aromatic L-amino acid decarboxylase (AAV2- hAADC) infusion into the brain
  Arms: VY-AADC02 (NBIb-1817)
Other: Sham (Placebo) Surgery — Bilateral partial burr/twist holes without dura penetration
  Arms: Sham (Placebo) Surgery

SUMMARY:
The objective of this study is to assess the safety of VY-AADC02 in participants with Parkinson's disease (PD) with motor fluctuations.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, 40 to 75 years of age (inclusive)
2. Diagnosis of PD, consistent with United Kingdom Brain Bank Criteria
3. Motor responsiveness to dopaminergic therapy, demonstrated by improvement in Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS III score)
4. Disease duration from diagnosis of ≥4 years
5. An average of ≥3 hours of OFF time (that is, periods of insufficient control of motor PD symptoms) per day over 3 consecutive days as confirmed by the PD Diary
6. A stable, optimal regimen of Parkinson's medications including levodopa for at least weeks prior to screening evaluation. Participants must have a minimum duration of levodopa treatment of ≥1 year
7. In the judgment of the Investigator, stable Parkinson's features and symptoms for at least 4 weeks prior to screening evaluation
8. Agrees to defer any elective neurological surgery, including deep brain stimulation or ablation procedure for PD, levodopa or apomorphine infusion, or the addition of new dopaminergic formulations until after the study is completed, if medically appropriate
9. Ability to travel to study visits

Key Exclusion Criteria:

1. Atypical or secondary parkinsonism, including but not limited to symptoms believed to be due to trauma, brain tumor, infection, cerebrovascular disease, other neurological disease, or to drugs, chemicals, or toxins, as determined by the Investigator
2. Montreal Cognitive Assessment (MoCA) score <26
3. New or unstable psychiatric conditions (psychosis, depression) within 1 year of screening
4. Brain imaging abnormalities in the striatum or other regions that would substantially increase risk of surgery
5. Contraindication to magnetic resonance imaging (MRI) and/or gadolinium-based contrast agents
6. Prior brain surgery, infusion therapies or planned treatments that could complicate the study procedure or negatively impact study evaluations as determined from participant interview, screening MRI, or medical records
7. History of malignancy other than treated carcinoma in situ within 3 years of screening evaluation
8. Prior gene transfer, current treatment with any investigational agent (drug or device) within 2 months of screening evaluation, or participation or plans to participate in another research study
9. Severe, biphasic and/or uncontrolled dyskinesia
10. Disabling or uncontrolled impulse control disorders

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (11):
- United States (11):
  - UC Irvine, Irvine, California
  - UC Davis Health System, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - NYU Langone Medical Center, New York, New York
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - University of Philadelphia, Dept of Neurology, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS: 1. GENE THERAPY FOR PARKINSON'S, 2. PHASE 3 STUDY IN FOCUS - INTEC PHARMA'S ACCORDION PILL, 3. CLINICAL TRIALS RESOURCES. J Parkinsons Dis. 2019;9(2):251-264. doi: 10.3233/JPD-199001. No abstract available. PMID 31127735